CLINICAL TRIAL: NCT04806828
Title: Preoperative Score of Inguinal Hernias. Is it Useful to Predict Outcomes
Acronym: POINTHER
Status: Completed | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, José A. Pereira, Consultat of Surgery, Hospital del Mar
Other Study IDs: POINTHER
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Inguinal Hernia
Keywords: Inguinal Hernia; Preoperative Score; Kingsnorth Score
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HF: Preoperative classification of inguinal hernia
  Interventions: Other: Preoperative classification

INTERVENTIONS:
Other: Preoperative classification — Score of inguinal hernia

SUMMARY:
To analyze and validate a preoperative score of difficulty of inguinal hernias and its correlation with postoperative outcomes

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age > 18 years
* Primary inguinal hernia
* Unilateral hernia
* Elective surgery

Exclusion Criteria:

* Recurrent inguinal hernia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inguinal hernia are more frequent in men and different characteristics
Study Population: All patients scheduled for a primary repair of inguinal hernia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  Rate of postoperative complications

SECONDARY OUTCOMES:
Lenght of operation | Intraoperative
  Minutes of operation
Recurrences | 1 year
  Recurrences during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pereira, Principal Investigator — Parc de Salut Mar
Locations (1):
- José Antonio Pereira, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No